CLINICAL TRIAL: NCT05138965
Title: Research About the Method of Cotton Padding Promoting the Healing of the Wound After Rectovaginal Fistula Surgery
Brief Title: the Method of Cotton Padding Promoting the Rectovaginal Fistula Surgery
Status: Completed | Type: Observational
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, FENG Li-peng, Attending Doctor, China Academy of Chinese Medical Sciences
Other Study IDs: 2021-11-15
Record Dates: First submitted 2021-11-15; First posted 2021-12-01 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Healing of the Wound After Rectovaginal Fistula Surgery
Keywords: Rectovaginal Fistula; Healing; Cotton Padding
MeSH Terms: conditions — Rectovaginal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- using the mCP: When the secretion reducing or the wound suture being removed, two pieces of 5cm×7cm-12p sterile gauzes will be crimped by the long side as the center of the reel,and be made as cylindrical gauze rolls with about D=1.5cm. After cleaning the wound, the cylindrical gauze rolls with its surface covered by alginates dressing will be placed above the vaginal wound with the help of endoscope.Itself tension of the rolls pressuring on the wound and the deep tissue can promote the wound healing. The rolls will be placed on about 5-6 hours every time, 2 times a day, for 7 days.Then observing the wound, if necessary, the method will be executed for another 7 days.
  Interventions: Procedure: the mCP with alginates dressing
- no using the mCP: When the secretion reducing or the wound suture bing removed, only alginates dressing will be placed above the vaginal wound with the help of endoscope, without any pressure, being placed about 5-6 hours every time, 2 times a day, for 7 days.
  Interventions: Procedure: only alginates dressing

INTERVENTIONS:
Procedure: the mCP with alginates dressing — The method is to use gauzes folded onto the RVF wound surface to compact the deep wound so as to solid and durable,when the gauzes surface will be covered by alginates dressing.
  Other Names: the method of cotton padding with alginates dressing
  Groups: using the mCP
Procedure: only alginates dressing — Only alginates dressing will be placed above the RVF wound without any pressure.
  Other Names: only alginates dressing without the mCP
  Groups: no using the mCP

SUMMARY:
The method of Cotton Padding (mCP) was summarized by combining with many years clinical experience and the traditional ancient books.The mCP could be used in Rectovaginal Fistula (RVF) post operation effectively,in order to improve the wound.The research aim is to observe if the mCP could influence the time of staying in hospital, healing time after RVF surgery.

DETAILED DESCRIPTION:
The method of Cotton Padding (mCP) originating from extensive and profound traditional chinese medicine (TCM) and being one of traditional surgical treatments of chronic wounds,could promote the wound healing after RVF surgery in previous clinical experience.

The research aim is to observe if the mCP could influence the time of staying in hospital, healing time,quality of life,complications after RVF surgery.

Also,investigators will try to explain the mechanism about the mDM improving the wound healing by the chinese architectural theory and the nanomechanical properties.

ELIGIBILITY:
Inclusion Criteria:

* rectovaginal fistula because of parturition,stapler,traumatic injury.

Exclusion Criteria:

* rectovaginal fistula because of IBD,radiation,cancer.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Rectovaginal fistulae are rare and account for less than 5% of all anorectal fistulae[1,2].
  The most common cause of RVF is obstetric trauma[2]. Trauma to the rectum, perineum,or vagina may cause RVF.The commonest form of trauma is during or following surgery, although blunt or penetrating trauma to the perineum or use of a foreign body in the vagina or rectum are well-recognized causes.The use of surgical stapling devices during stapled hemorrhoidectomy and stapled transanal rectal resections (STARR) have been implicated.
  (© Springer Nature Switzerland AG 2021. G.A.Santoro et al. (eds.), Pelvic Floor Disorders, https://doi.org/10.1007/978-3-030-40862-6_79)
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
the time of healing | 28days-40days
  the time of healing

SECONDARY OUTCOMES:
the time of staying hospital | 7days-21days
  the time of staying hospital
occurrence rate of complications | 1day-90days
  occurrence rate of complications,including recurrence,blooding,wound dehiscence.

OTHER OUTCOMES:
the quality of life post-operation | 90days-180days
  using the Wexner continence score (WCS) or the Vaizey score (VS) to assess the fecal incontinence,and using the Female sexual function index (FSFI) to assess the sex life,and aslo using the Clavien-Dindo classification(CDC) to assess other situation postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: LI guodong, Study Director — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (3):
- China (3):
  - Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing
  - Beijing Mayinglong Changqing Anorectal Hospital, Beijing
  - Southern District of Guang'an men Hospital,China Academy of Chinese Medical Sciences, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in the article after identification, excluding the private information of participants.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Becoming available after publication and ending 12 months following article publication.
Access Criteria: Proposals should be emailed to venus59514@sina.com.To gain access, data requestors will need to sign a data access agreement and offer payment.